CLINICAL TRIAL: NCT01332955
Title: Pilot Study of PegInterferon-Ribavirin-Telaprevir Efficacy and Tolerability in HIV-HCV Coinfected Patients Who Had Previously Failed a PegInterferon-Ribavirin Regimen. (ANRS HC26 TelapreVIH)
Brief Title: Telaprevir in HIV-HCV Coinfected Patients Who Had Previously Failed a Peginterferon-Ribavirin Regimen
Acronym: TelapreVIH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023287-41; ANRS HC26 TelapreVIH (Other: (Inserm-ANRS))
Record Dates: First submitted 2011-03-28; First posted 2011-04-11 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic; HIV Infection
Keywords: Hepatitis C, Chronic; HIV Infection; Telaprevir; Peginterferon alfa-2a; Ribavirin; Pharmacokinetic; Pharmacogenetic; Previous peginterferon-ribavirin regimen failure
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telaprevir-pegIFN alfa-2a-ribavirine (Experimental): Single Group Assignment
  Interventions: Drug: Telaprevir; Biological: pegIFN alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Drug : telaprevir, Tablet, Oral, 750 mg, q8h, 12 weeks if associated with atazanavir or raltegravir
  Drug : telaprevir, Tablet, Oral, 1125 mg, q8h, 12 weeks if associated with efavirenz
  Other Names: VX-950
Biological: pegIFN alfa-2a — Subcutaneous injection, 180 μg, once weekly, 48 weeks or 72 weeks
  Other Names: peginterferon alfa-2a, Pegasys®
Drug: Ribavirin — (weight-based dose) Tablet, Oral, 1000 mg for subjects weighing below 75 kg or 1200 mg for subjects weighing equal or over75 kg, once daily, 48 weeks or 72 weeks
  Other Names: Copegus®; Rebetol®

SUMMARY:
This phase II, multicentric, national pilot trial is designed to estimate the sustained virological response rate (SVR) following a 12 weeks treatment by telaprevir combined with a 48 or 72 weeks treatment by peginterferon and ribavirin, based upon the rapid virological response (RVR) at week 8 (4 weeks after telaprevir start), and to compare the observed SVR to 20%, a rate determining a significant therapeutic benefit in this population of patients. The primary endpoint will be the SVR defined as undetectable HCV-RNA measured 24 weeks after the end of therapy (EOT).

DETAILED DESCRIPTION:
This phase II pilot trial is designed for HIV-1 and HCV genotype 1 coinfected patients who had previously failed a peginterferon-ribavirin regimen.

Intervention Design:

* Induction, Lead-in, phase: day 0 to week 4 PegInterferon alpha-2a, 180 µg subcutaneous injection, once weekly + Ribavirin (weight-based dose) 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d.
* Telaprevir phase: week 4 to week 16 PegInterferon alpha-2a, 180 µg subcutaneous injection, once weekly + Ribavirin (weight-based dose) 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d.

  + Telaprevir 750 mg q 8h (or 1125 mg q 8h in association with Efavirenz)
* Maintenance phase: week 16 to week 48 or 72 PegInterferon alpha-2a, 180 µg subcutaneous injection, once weekly + Ribavirin (weight-based dose) 1000 mg for subjects weighing <75 kg or 1200 mg for subjects weighing ≥75 kg, b.i.d.

The duration of the maintenance phase is determined by the RVR at week 8 (4 weeks after Telaprevir start.

Complete RVR (not measurable HCV-RNA at week 8): maintenance from week 16 to week 48

_Partial RVR (HCV-RNA below 1 000 UI/mL but still measurable at week 8): maintenance phase from week 16 to week 48

And stable antiretroviral treatment for over 3 months among the authorized combinations: (tenofovir 300 mg, emtricitabine 200 mg, atazanavir 300 mg, ritonavir 100 mg) q.d. or (tenofovir 300 mg, emtricitabine 200 mg, efavirenz 600 mg) q.d. or (tenofovir 300 mg, emtricitabine 200 mg q.d. and raltegravir 400 mg b.i.d.) once Drug-Drug interaction data will be available. Patients who could not receive one of these 3 combinations can be included if they are receiving a stable combination of at least 3 drugs among the following: tenofovir, emtricitabine/lamivudine, efavirenz, atazanavir-boosted or not, raltegravir (once Drug-Drug interaction data will be available). These patients cannot participate in the pharmacokinetic study.

The trial will enroll 80 subjects. The proportion of patients included, presenting with cirrhosis (METAVIR F4) will remain below 50% of all patients The proportion of patients included, null-responders to previous HCV treatment (HCV-RNA decline at week 12 less than 2 log10 UI/ml) but no cirrhosis (maximum equal METAVIR F3) will remain below 30% of patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed at screening visit at the latest
* Patient registered with or covered by a social security scheme
* HIV-1 infection
* Chronic, genotype 1, hepatitis C with detectable HCV RNA at screening
* Virological failure following a previous treatment of at least 12 weeks by peginterferon alpha-2a ≥ 135 µg once weekly or peginterferon alpha-2b ≥ 1.0 µg per kg once weekly + ribavirin ≥ 600 mg once daily. Virological failure defined by persistence of a detectable HCV-RNA, with the same genotype than before. Null responder patient, with less than 2 Log10 HCV-RNA decline at week 12 with cirrhosis are excluded from the study. Null responder patients without cirrhosis (equal or below METAVIR F3) are limited to less than 30 % of all patients included
* No Interferon and/or Ribavirin within past 6 months
* Stable antiretroviral treatment for over 3 months at screening. Authorized combinations: tenofovir-emtricitabine-boosted atazanavir,tenofovir-emtricitabine-efavirenz,tenofovir-emtricitabine-raltegravir, once Drug-Drug interaction data will be available. Patients with a stable combination of at least 3 of the following drugs: tenofovir, emtricitabine/lamivudine, efavirenz, atazanavir-boosted or not, raltegravir. These patients cannot participate in the pharmacokinetic study
* CD4 >200/mm3 and >15% at screening
* Plasma HIV-RNA <50 copies/mL for at least 6 months at screening visit
* Body weight ≥ 40 kg to equal or below 125 kg
* Fibrosis stage have to be documented by a significant liver biopsy (cumulative length ≥ 15 mm or ≥ 6 portal spaces), within 3 years. Patients with a previous liver biopsy exhibiting cirrhosis lesions (METAVIR F4) are allowed to enter the study without a new biopsy. The proportion of patients with cirrhosis lesions (METAVIR F4) is limited to 50% of all patients.
* Male patients, female patients with child-bearing potency and their heterosexual partners must use an adequate contraception from 1 month before initiation of treatment to 7 months following the end of treatment for men and to 4 months following the end of treatment for women. Subjects (or their female partners) must not be pregnant or planning to become pregnant within 2 years after enrolling in the study

Exclusion Criteria:

* Patient with liver failure (Child B and C) or past history of decompensated cirrhosis
* Significant oesophageal varices (Stages 2-3) on a gastrointestinal endoscopy within 3 years
* Detectable AgHBs
* HIV-2 co-infection
* Contra-indication to ribavirin or peginterferon
* Severe pre-existing cardiac or pulmonary disease
* Untreated dysthyroidism
* Uncontrolled Type 2 diabetes
* Optic neuritis past history and retinal condition
* History of organ transplant
* Severe hemoglobinopathy
* Congenital QT prolongation, family history of congenital QT prolongation or sudden unexpected death
* Contra-indication to telaprevir, hypersensitivity to any component of the drug product
* Any disease requiring long term, systemic corticotherapy or immunosuppressive therapy during study
* Alcohol intake that may represent an obstacle for the participation of the subject
* Substance abuse that may represent an obstacle for the participation of the subject
* Acute CDC stage C opportunistic infection within the previous 6 months
* Past history of cancer within the previous 5 years (except skin basal cell carcinoma, Kaposi's disease in stable remission, in situ cervical cancer and in situ anal cancer)
* Any active malignant disease including hepatocellular carcinoma
* Patients unable to observe the study procedures
* Participation to another clinical trial within the previous 30 days
* Haemoglobin <120 g/L for women and <130 g/L for men
* Platelets <90 000/mm3
* Neutrophils <1 500/mm3
* Renal insufficiency defined by an estimated Glomerular Filtration Rate < 60 mL/mn (MDRD equation)
* Associated medication susceptible to interfere with the pharmacokinetic parameters of telaprevir and/or antiretroviral associated drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Estimation of SVR following a 12 wks treatment by telaprevir combined with a 48 or 72 wks peginterferon-ribavirin treatment, based upon the rapid virological response, and comparison to 20% (which would correspond to a significant therapeutic benefit) | up to 92 weeks or 116 weeks depending on rapid virologic response
  HCV-RNA measured 24 weeks after the end of HCV treatment

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From week 0 up to 92 weeks or 116 weeks depending on rapid virologic response
Estimation of the Sustained Virological Response defined as undetectable HCV-RNA at Week 12 after the end of HCV treatment | at Week 60 or Week 84 depending on rapid virologic response
  HCV-RNA measured 12 weeks after the end of HCV treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent COTTE, MD, Principal Investigator — Hopital Croix Rousse LYON FRANCE; Jean-Pierre ABOULKER, MD, Study Chair — INSERM SC10 VILLEJUIF FRANCE
Locations (1):
- Service Maladies Infectieuses et Tropicales, Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Derived] Cotte L, Braun J, Lascoux-Combe C, Vincent C, Valantin MA, Sogni P, Lacombe K, Neau D, Aumaitre H, Batisse D, de Truchis P, Gervais A, Michelet C, Morlat P, Vittecoq D, Rosa I, Bertucci I, Chevaliez S, Aboulker JP, Molina JM; French National Agency for Research on AIDS and Viral Hepatitis (ANRS) HC26 Study Group. Telaprevir for HIV/hepatitis C virus-coinfected patients failing treatment with pegylated interferon/ribavirin (ANRS HC26 TelapreVIH): an open-label, single-arm, phase 2 trial. Clin Infect Dis. 2014 Dec 15;59(12):1768-76. doi: 10.1093/cid/ciu659. Epub 2014 Aug 18. PMID 25139963
- See also: Related Info — http://www.anrs.fr